CLINICAL TRIAL: NCT06402552
Title: A Randomized Controlled Trial Comparing Bp-MRI and Mp-MRI on the Screening Accuracy for Clinically Significant Prostate Cancer Before MRI-fusion Targeted Biopsy
Brief Title: Comparing Bp-MRI and Mp-MRI for Prostate Cancer Screening Accuracy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202400317A3
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Randomized Controlled Trial; Prostate Cancer; Magnetic Resonance Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prostate cancer (Experimental): Patients who are suspicious of prostate cancers with abnormal digital examination, or abnormal ultrasound and having a pre-MRI and were scheduled to receive prostate biopsy will be enrolled in this study. Patients will be randomized in a 1:1 manner to bp-MRI and mp-MRI. Patients with clinical suspicion of prostate cancer on MRI with PI-RADS (Prostate Imaging-Reporting and Data System, version 2.1)
  Interventions: Diagnostic Test: bp-MRI prostate; Diagnostic Test: mp-MRI prostate

INTERVENTIONS:
Diagnostic Test: bp-MRI prostate — Biparametric MRI is considered less comprehensive compared to multiparametric MRI (mp-MRI), which includes additional parameters like dynamic contrast-enhanced MRI (DCE-MRI). However, bp-MRI offers a simpler, faster, and often less expensive alternative that still provides critical diagnostic information, particularly in the detection of clinically significant prostate cancer. It's commonly used where less comprehensive assessment is sufficient or in situations where contrast use is contraindicated.
Diagnostic Test: mp-MRI prostate — Multiparametric MRI is highly valued for its ability to improve the detection and characterization of clinically significant prostate cancer, aid in biopsy guidance, and help in treatment planning and monitoring. Its comprehensive approach provides crucial insights that are not as readily available through simpler imaging modalities like biparametric MRI (bp-MRI).

SUMMARY:
3.1 Study Objectives: 3.1.1 Primary objective: The investigators aim to address these questions for Taiwan males suspicious of csPCA, with PSA range of 4-20 ng/ml by conducting a RCT trial.

3.2 Study endpoints: 3.2.1 Primary endpoint: The proportion of men with clinically significant Prostate cancer(csPCa), defined as a diagnosis of ISUP (International Society of Urogenital Pathology) Grade group ≥2 prostate cancer, in at least one biopsy core.

3.2.2 Secondary endpoints:

1. The proportion of men with a diagnosis of any PCa
2. The proportion of men with a diagnosis of clinically insignificant PCa, defined as ISUP grade group 1 PCa (ISUP 1 PCa)
3. The proportion of men with a diagnosis of csPCa
4. Only in targeted biopsy
5. Only in systematic biopsy
6. The proportion of csPCa of all suspicious lesions from bp-MRI and mp-MRI.

DETAILED DESCRIPTION:
Study intervention MRI prostate Bi-parametric and multi-parametric MRI prostates can be performed using a 3.0 Tesla scanner with a pelvic phased array coil with or without contrast. MRI findings will be reported according to PI-RADS (Prostate Imaging-Reporting and Data Systems) v2.1 recommendations. MRI will be reported by radiologists with experience in MRI prostate reporting. PI-RADS scores 3-5 will be regarded as suspicious, and targeted plus systematic biopsy will be performed.

Prostate biopsy In patients with suspicious lesion found on MRI (identified as PI-RADS score 3-5 lesions on bp-MRI or mp-MRI), biopsies will be done via trans-perineal approach under general anesthesia with 3 cores of targeted biopsy from each lesion, alone with 3 cores of systemic biopsy from right and left lobes respectively.

In those without identified suspicious lesions on MRI, a standard 12-core systematic biopsy will be performed via trans-rectal approach under local anesthesia.

All biopsies will be performed by Urologists experienced in both targeted and systemic prostate biopsy. Targeted biopsies will be done by software-assisted MRI-USG fusion registration. Peri-biopsy antibiotics are given according to our clinical guidelines.

Post-biopsy management Patients will be discharged after prostate biopsy when they can pass urine without significant gross hematuria, and clinically stable. They will be followed up in the clinic within 10 days after a biopsy to review pathology results and complications. All biopsies will be assessed by experienced Urogenital pathologists and reported according to the International Society of Urological Pathology (ISUP) consensus. The study period ends after the first clinic follow-up.

In our medical research, the investigators prioritize protecting participant privacy and confidentiality. The investigators use unique research codes to anonymize personal details like names and IDs. The principal investigator keeps consultation results and diagnoses confidential, even in published research. Participants consent to have their records reviewed by authorized parties for legal and ethical compliance, with a promise of maintaining their anonymity. For safety, the investigators may inform participants' other doctors about their trial involvement to manage treatment interactions. Overall, these steps ensure participant privacy and safety throughout the research.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥50 years of age
2. Clinical suspicion of prostate cancer and indicated for prostate biopsy
3. Serum Prostate-specific antigen (PSA) between 4~20 ng/mL
4. Eligible for MRI study
5. Digital rectal examination ≤ cT2 (organ-confined cancer)
6. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy in the 6 months before screening visit
2. Prior diagnosis of prostate cancer
3. Contraindicated to prostate biopsy: active urinary tract infection, failed insertion of transrectal ultrasound probe into rectum (abdominal perineal resection, anal stenosis), uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped (continue low-dose aspirin before and after biopsy is permitted)
4. Contraindicated to MRI study: contrast medium allergy, claustrophobia, or other contraindications (e.g.: intra-abdominal metal foreign bodies).
5. Patients without histological results of prostate biopsies due to patient refusal for biopsy or loss of follow up before biopsy being done
6. Patients have prior treatments for prostate cancers or any kinds of hormone therapy, immunotherapy, chemotherapy, radiation therapy of the pelvic cavity.
7. Patients' withdrawal of informed consents of this study

Withdrawal criteria:

1. Patients could not complete the scheduled MRI examinations
2. MRI images of insufficient quality to localized csPCA or to exclude the presence of csPCA

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient only
Enrollment: 370 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Clinically Significant Prostate Cancer among Men as Defined by ISUP Grade Group ≥2 in Biopsy Samples | 2-3 weeks
  The proportion of men with clinically significant Prostate cancer(csPCa), defined as a diagnosis of ISUP (International Society of Urogenital Pathology) Grade group ≥2 prostate cancer, in at least one biopsy core.

SECONDARY OUTCOMES:
Prostate Cancer Diagnosis Rates and Specifics in Biopsy Methods | 4-6 weeks
  1. The proportion of men with a diagnosis of any PCa
  2. The proportion of men with a diagnosis of clinically insignificant PCa, defined as ISUP grade group 1 PCa (ISUP 1 PCa)
  3. The proportion of men with a diagnosis of csPCa
  4. Only in targeted biopsy
  5. Only in systematic biopsy
  6. The proportion of csPCa of all suspicious lesions from bp-MRI and mp-MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan, Taiwan

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT06402552/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT06402552/ICF_001.pdf